CLINICAL TRIAL: NCT01165203
Title: Safety and Immunogenicity of GlaxoSmithKline Biologicals' Herpes Zoster Vaccine 1437173A in Adult HIV-infected Subjects
Brief Title: Study to Evaluate GSK Biologicals' Herpes Zoster Vaccine GSK1437173A in Human Immunodeficiency Virus (HIV)-Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112673
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2017-10

CONDITIONS: Herpes Zoster
Keywords: immunogenicity; vaccine; safety; HIV; Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- GSK1437173A Group (Experimental): Subjects who received three doses of GSK1437173A vaccine (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Herpes Zoster Vaccine GSK1437173A
- Placebo Group (Placebo Comparator): Subjects who received three doses of placebo (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes Zoster Vaccine GSK1437173A — intramuscular injection
  Other Names: HZ/su vaccine
  Arms: GSK1437173A Group
Biological: Placebo — intramuscular injection
  Arms: Placebo Group

SUMMARY:
This observer-blind study will evaluate the safety and immunogenicity of GlaxoSmithKline (GSK) Biologicals' investigational Herpes Zoster (HZ) vaccine GSK1437173A in Human Immunodeficiency Virus (HIV) infected subjects, firstly enrolling subjects treated with antiretroviral therapy (ART) and with high CD4 T cell counts, and subsequently ART-treated subjects with low CD4 T cell counts, and ART-naïve subjects with high CD4 T cell counts.

This Protocol Posting has been updated following Amendment 1 of the Protocol, August 2010. The impacted sections is exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol;
* Male and female subjects at least 18 years old at the time of vaccination;
* Subjects born before 1985 and not from a tropical region. Subjects born in 1985 or later and subjects born before 1985 in tropical regions must have a history of Varicella Zoster virus (VZV) infection or serological evidence of prior VZV infection;
* Written informed consent obtained from the subject;
* Female subjects of non-childbearing potential may be enrolled in the study; Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.

OR Female subjects of childbearing potential may be enrolled in the study, if the subject has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series;

* Known to be human immunodeficiency virus-1 (HIV-1) infected, diagnosed at least 1 year prior to enrolment;
* For the antiretroviral therapyART High CD4 and ART Low CD4 cohorts:

  * Stable on ART for at least one year
  * CD4 T cell count >= 50 cells /mm3 at screening
  * Undetectable VL at screening;
* For the non-ART High CD4 cohort:

  * ART-naïve subjects who have never received anti-retroviral therapy after HIV diagnosis and for whom commencement of ART is not expected based on current assessment within next seven months;
  * HIV VL >= 1000 copies/mL and <= 100 000 copies/mL at screening
  * CD4 T cell count >= 500 cells/mm3 at screening.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period;
* Vaccination against varicella or herpes zoster (HZ) within the previous 12 months;
* Occurrence of a varicella or HZ episode within the previous 12 months;
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Additionally, consider allergic reactions to other material or equipment related to study participation. Please note, the vaccine and vials in this study do not contain latex;
* Has currently an Acquired Immunodeficiency Syndrome (AIDS) defining condition;
* Opportunistic infection or AIDS-associated malignancy in the previous year;
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease other than HIV infection or immunosuppressive/cytotoxic therapy;
* Administration of immunoglobulins, and/or any blood products within 90 days preceding the first dose of study vaccine/placebo or planned administration during the study period;
* Chronic administration of immunosuppressive or other immune-modifying drugs within 6 months prior to the first vaccine dose;
* Administration and/or planned administration of a vaccine not foreseen by the study protocol within 30 days before dose 1, dose 2 and/or 3 of vaccine and/or within 30 days after any dose. However, licensed non-replicating vaccines may be administered up to 8 days prior to dose 1, 2 and/or 3, and/or at least 14 days after any dose of study vaccine;
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product;
* Acute disease at the time of enrolment;
* Any contraindication to receiving intramuscular injections;
* Any condition or illness which might interfere with the evaluation of the safety or immunogenicity of the vaccine;
* Active hepatitis B (HBV) infection or active hepatitis C (HCV) infection.
* Current use of HIV fusion inhibitors, chemokine (C-C motif) receptor (CCR5) inhibitors or Interleukin-2/ Interleukin-7/ Interferon;
* For subjects in the ART cohorts, any change in anti-retroviral drug regimen within 12 weeks prior to vaccination;
* Pregnant or lactating female;
* Female planning to become pregnant or planning to discontinue contraceptive precautions;
* Abnormal biochemical and hematological laboratory values obtained for blood samples collected at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2012-07-06 (Actual); Study Completion 2013-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (5):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Santa Fe, New Mexico
  - GSK Investigational Site, Dallas, Texas
- Germany (6):
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- United Kingdom (2):
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Berkowitz EM, Moyle G, Stellbrink HJ, Schurmann D, Kegg S, Stoll M, El Idrissi M, Oostvogels L, Heineman TC; Zoster-015 HZ/su Study Group. Safety and immunogenicity of an adjuvanted herpes zoster subunit candidate vaccine in HIV-infected adults: a phase 1/2a randomized, placebo-controlled study. J Infect Dis. 2015 Apr 15;211(8):1279-87. doi: 10.1093/infdis/jiu606. Epub 2014 Nov 3. PMID 25371534
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112673 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Active Phase
Arm/Group | GSK1437173A Group | Placebo Group
Started | 74 | 49
Completed | 69 | 47
Not Completed | 5 | 2
Not completed — Serious Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Migrated/moved from study area | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Period: Extended Safety Follow-up Phase
Arm/Group | GSK1437173A Group | Placebo Group
Started | 74 | 49
Completed | 67 | 45
Not Completed | 7 | 4
Not completed — Serious Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Migrated/moved from study area | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other-subjects business reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1437173A Group | Placebo Group | Total
Number analyzed (Participants) | 74 | 49 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (10.68) | 45.1 (11.36) | 46.0 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 69 | 47 | 116
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 6 | 2 | 8
  Asian-East Asian heritage | 0 | 1 | 1
  Asian-Japanese heritage | 1 | 0 | 1
  White-Caucasian/European heritage | 66 | 42 | 108
  Unspecified | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 18
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants | 6 | 2

2. Primary Outcome: Number of Subjects With SAEs Related to Study Participation or to a Concurrent GSK Medication/Vaccine
Description: as for outcome 1
Time Frame: From screening (up to 21 days prior to Month 0) until Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants | 0 | 0

3. Primary Outcome: Number of Subjects With Any Fatal SAEs
Description: as for outcome 1
Time Frame: From screening (up to 21 days prior to Month 0) until Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants | 0 | 0

4. Primary Outcome: Number of Subjects With Any Adverse Events (AEs) of Specific Interest
Description: AEs of specific interest include new onset of autoimmune diseases (NOADs) and other immune mediated inflammatory disorders from administration of the first dose of vaccine/placebo.
Time Frame: From Month 0 until Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- GSK1437173A Group: Subjects who received three doses of gE/AS01B vaccine (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants | 0 | 0

5. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = incidence of a particular symptom regardless of their intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 73 | 48
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 72 | 48
  Any Pain, Dose 1 | 69 | 4
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Pain, Dose 1 | 4 | 0
  Any Redness, Dose 1: number analyzed (Participants) | 72 | 48
  Any Redness, Dose 1 | 17 | 0
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Redness, Dose 1 | 2 | 0
  Any Swelling, Dose 1: number analyzed (Participants) | 72 | 48
  Any Swelling, Dose 1 | 12 | 0
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Swelling, Dose 1 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 66 | 44
  Any Pain, Dose 2 | 57 | 3
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Pain, Dose 2 | 8 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 66 | 44
  Any Redness, Dose 2 | 19 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 66 | 44
  Any Swelling, Dose 2 | 11 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 53 | 38
  Any Pain, Dose 3 | 43 | 1
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Pain, Dose 3 | 7 | 0
  Any Redness, Dose 3: number analyzed (Participants) | 53 | 38
  Any Redness, Dose 3 | 9 | 0
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Redness, Dose 3 | 2 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 53 | 38
  Any Swelling, Dose 3 | 5 | 0
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Swelling, Dose 3 | 0 | 0
  Any Pain, Across doses | 72 | 6
  Grade 3 Pain, Across doses | 12 | 0
  Any Redness, Across doses | 28 | 0
  Grade 3 Redness, Across doses | 4 | 0
  Any Swelling, Across doses | 20 | 0
  Grade 3 Swelling, Across doses | 1 | 0

6. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal (symptoms included nausea, vomiting, diarrhoea and/or abdominal pain), headache, myalgia, shivering and temperature [defined as oral/axillary temperature above (>) 37.5 degrees Celsius (°C)]. Any = incidence of a particular symptom regardless of their intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 73 | 48
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 72 | 48
  Any Fatigue, Dose 1 | 30 | 13
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Fatigue, Dose 1 | 0 | 3
  Related Fatigue, Dose 1: number analyzed (Participants) | 72 | 48
  Related Fatigue, Dose 1 | 17 | 8
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 72 | 48
  Any Gastrointestinal, Dose 1 | 13 | 8
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 72 | 48
  Related Gastrointestinal, Dose 1 | 6 | 6
  Any Headache, Dose 1: number analyzed (Participants) | 72 | 48
  Any Headache, Dose 1 | 25 | 10
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Headache, Dose 1 | 0 | 1
  Related Headache, Dose 1: number analyzed (Participants) | 72 | 48
  Related Headache, Dose 1 | 16 | 6
  Any Myalgia, Dose 1: number analyzed (Participants) | 72 | 48
  Any Myalgia, Dose 1 | 34 | 6
  Grade 3 Myalgia, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Myalgia, Dose 1 | 4 | 0
  Related Myalgia, Dose 1: number analyzed (Participants) | 72 | 48
  Related Myalgia, Dose 1 | 26 | 6
  Any Shivering, Dose 1: number analyzed (Participants) | 72 | 48
  Any Shivering, Dose 1 | 19 | 5
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Shivering, Dose 1 | 0 | 0
  Related Shivering, Dose 1: number analyzed (Participants) | 72 | 48
  Related Shivering, Dose 1 | 11 | 5
  Any Temperature, Dose 1: number analyzed (Participants) | 72 | 48
  Any Temperature, Dose 1 | 7 | 2
  Grade 3 Temperature, Dose 1: number analyzed (Participants) | 72 | 48
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1: number analyzed (Participants) | 72 | 48
  Related Temperature, Dose 1 | 2 | 2
  Any Fatigue, Dose 2: number analyzed (Participants) | 66 | 44
  Any Fatigue, Dose 2 | 41 | 8
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Fatigue, Dose 2 | 7 | 3
  Related Fatigue, Dose 2: number analyzed (Participants) | 66 | 44
  Related Fatigue, Dose 2 | 25 | 5
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 66 | 44
  Any Gastrointestinal, Dose 2 | 18 | 3
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Gastrointestinal, Dose 2 | 1 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 66 | 44
  Related Gastrointestinal, Dose 2 | 8 | 1
  Any Headache, Dose 2: number analyzed (Participants) | 66 | 44
  Any Headache, Dose 2 | 32 | 3
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Headache, Dose 2 | 3 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 66 | 44
  Related Headache, Dose 2 | 18 | 1
  Any Myalgia, Dose 2: number analyzed (Participants) | 66 | 44
  Any Myalgia, Dose 2 | 33 | 4
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Myalgia, Dose 2 | 1 | 1
  Related Myalgia, Dose 2: number analyzed (Participants) | 66 | 44
  Related Myalgia, Dose 2 | 24 | 2
  Any Shivering, Dose 2: number analyzed (Participants) | 66 | 44
  Any Shivering, Dose 2 | 23 | 1
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Shivering, Dose 2 | 4 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 66 | 44
  Related Shivering, Dose 2 | 17 | 1
  Any Temperature, Dose 2: number analyzed (Participants) | 66 | 44
  Any Temperature, Dose 2 | 12 | 1
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 66 | 44
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 66 | 44
  Related Temperature, Dose 2 | 10 | 0
  Any Fatigue, Dose 3: number analyzed (Participants) | 53 | 38
  Any Fatigue, Dose 3 | 36 | 6
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Fatigue, Dose 3 | 7 | 1
  Related Fatigue, Dose 3: number analyzed (Participants) | 53 | 38
  Related Fatigue, Dose 3 | 24 | 3
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 53 | 38
  Any Gastrointestinal, Dose 3 | 8 | 4
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Gastrointestinal, Dose 3 | 1 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 53 | 38
  Related Gastrointestinal, Dose 3 | 5 | 2
  Any Headache, Dose 3: number analyzed (Participants) | 53 | 38
  Any Headache, Dose 3 | 33 | 7
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Headache, Dose 3 | 4 | 1
  Related Headache, Dose 3: number analyzed (Participants) | 53 | 38
  Related Headache, Dose 3 | 21 | 3
  Any Myalgia, Dose 3: number analyzed (Participants) | 53 | 38
  Any Myalgia, Dose 3 | 32 | 1
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Myalgia, Dose 3 | 6 | 0
  Related Myalgia, Dose 3: number analyzed (Participants) | 53 | 38
  Related Myalgia, Dose 3 | 22 | 1
  Any Shivering, Dose 3: number analyzed (Participants) | 53 | 38
  Any Shivering, Dose 3 | 20 | 1
  Grade 3 Shivering, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Shivering, Dose 3 | 7 | 0
  Related Shivering, Dose 3: number analyzed (Participants) | 53 | 38
  Related Shivering, Dose 3 | 14 | 1
  Any Temperature, Dose 3: number analyzed (Participants) | 53 | 38
  Any Temperature, Dose 3 | 11 | 1
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 53 | 38
  Grade 3 Temperature, Dose 3 | 0 | 0
  Related Temperature, Dose 3: number analyzed (Participants) | 53 | 38
  Related Temperature, Dose 3 | 6 | 0
  Any Fatigue, Across doses | 55 | 14
  Grade 3 Fatigue, Across doses | 12 | 4
  Related Fatigue, Across doses | 41 | 8
  Any Gastrointestinal, Across doses | 28 | 11
  Grade 3 Gastrointestinal, Across doses | 2 | 1
  Related Gastrointestinal, Across doses | 16 | 7
  Any Headache, Across doses | 47 | 15
  Grade 3 Headache, Across doses | 6 | 2
  Related Headache, Across doses | 34 | 8
  Any Myalgia, Across doses | 54 | 9
  Grade 3 Myalgia, Across doses | 10 | 1
  Related Myalgia, Across doses | 44 | 8
  Any Shivering, Across doses | 37 | 5
  Grade 3 Shivering, Across doses | 11 | 0
  Related Shivering, Across doses | 29 | 5
  Any Temperature, Across doses | 22 | 3
  Grade 3 Temperature, Across doses | 0 | 0
  Related Temperature, Across doses | 17 | 2

7. Primary Outcome: Number of Subjects With Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days (Days 0-29) after each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants
  Any AE(s) | 41 | 26
  Grade 3 AE(s) | 4 | 2
  Related AE(s) | 11 | 3

8. Primary Outcome: Number of Subjects With Any Hematological and Biochemical Parameters Below, Within or Above Normal Laboratory Ranges
Description: The assessed parameters were Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Basophils, Bilirubin Total, Bilirubin Conjugated / Direct, Creatinine, Eosinophils, Glucose, Bicarbonate, Haemoglobin, Potassium, Lymphocytes, Monocytes, Sodium, Neutrophils, Platelets and White Blood Cells. Tabulation was made by relation to the normal laboratory ranges: below, within or above, and also status unknown.
Time Frame: At Screening Visit (up to 21 days prior to Month 0)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants
  Alanine Aminotransferase: Unknown | 0 | 0
  Alanine Aminotransferase: Below | 0 | 0
  Alanine Aminotransferase: Within | 70 | 41
  Alanine Aminotransferase: Above | 4 | 8
  Albumin: Unknown | 0 | 0
  Albumin: Below | 0 | 0
  Albumin: Within | 72 | 47
  Albumin: Above | 2 | 2
  Alkaline Phosphatase: Unknown | 0 | 0
  Alkaline Phosphatase: Below | 0 | 0
  Alkaline Phosphatase: Within | 70 | 44
  Alkaline Phosphatase: Above | 4 | 5
  Aspartate Aminotransferase: Unknown | 0 | 0
  Aspartate Aminotransferase: Below | 0 | 0
  Aspartate Aminotransferase: Within | 69 | 45
  Aspartate Aminotransferase: Above | 5 | 4
  Basophils: Unknown | 0 | 0
  Basophils: Below | 0 | 0
  Basophils: Within | 74 | 49
  Basophils: Above | 0 | 0
  White Blood Cells: Unknown | 1 | 0
  White Blood Cells: Below | 3 | 0
  White Blood Cells: Within | 69 | 47
  White Blood Cells: Above | 1 | 2
  Total Bilirubin: Unknown | 0 | 0
  Total Bilirubin: Below | 0 | 0
  Total Bilirubin: Within | 65 | 46
  Total Bilirubin: Above | 9 | 3
  Bilirubin Conjugated / Direct: Unknown | 0 | 0
  Bilirubin Conjugated / Direct: Below | 0 | 0
  Bilirubin Conjugated / Direct: Within | 73 | 49
  Bilirubin Conjugated / Direct: Above | 1 | 0
  Creatinine: Unknown | 0 | 0
  Creatinine: Below | 6 | 8
  Creatinine: Within | 68 | 40
  Creatinine: Above | 0 | 1
  Eosinophils: Unknown | 0 | 0
  Eosinophils: Below | 14 | 10
  Eosinophils: Within | 59 | 38
  Eosinophils: Above | 1 | 1
  Glucose: Unknown | 0 | 0
  Glucose: Below | 0 | 1
  Glucose: Within | 69 | 43
  Glucose: Above | 5 | 5
  Bicarbonate: Unknown | 0 | 0
  Bicarbonate: Below | 5 | 2
  Bicarbonate: Within | 69 | 47
  Bicarbonate: Above | 0 | 0
  Haemoglobin: Unknown | 0 | 0
  Haemoglobin: Below | 13 | 5
  Haemoglobin: Within | 58 | 42
  Haemoglobin: Above | 3 | 2
  Potassium: Unknown | 0 | 0
  Potassium: Below | 0 | 0
  Potassium: Within | 74 | 49
  Potassium: Above | 0 | 0
  Lymphocytes: Unknown | 0 | 0
  Lymphocytes: Below | 0 | 1
  Lymphocytes: Within | 74 | 48
  Lymphocytes: Above | 0 | 0
  Monocytes: Unknown | 0 | 0
  Monocytes: Below | 2 | 4
  Monocytes: Within | 71 | 45
  Monocytes: Above | 1 | 0
  Sodium: Unknown | 0 | 0
  Sodium: Below | 1 | 0
  Sodium: Within | 73 | 49
  Sodium: Above | 0 | 0
  Neutrophils: Unknown | 0 | 0
  Neutrophils: Below | 5 | 3
  Neutrophils: Within | 69 | 45
  Neutrophils: Above | 0 | 1
  Platelets: Unknown | 0 | 0
  Platelets: Below | 4 | 1
  Platelets: Within | 70 | 48
  Platelets: Above | 0 | 0

9. Primary Outcome: Number of Subjects With Any Hematological and Biochemical Parameters Below, Within or Above Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 73 | 45
Participants
  Alanine Aminotransferase: Unknown | 0 | 0
  Alanine Aminotransferase: Below | 0 | 0
  Alanine Aminotransferase: Within | 67 | 41
  Alanine Aminotransferase: Above | 6 | 4
  Albumin: Unknown | 0 | 0
  Albumin: Below | 0 | 0
  Albumin: Within | 69 | 43
  Albumin: Above | 4 | 2
  Alkaline Phosphatase: Unknown | 0 | 0
  Alkaline Phosphatase: Below | 0 | 0
  Alkaline Phosphatase: Within | 71 | 43
  Alkaline Phosphatase: Above | 2 | 2
  Aspartate Aminotransferase: Unknown | 0 | 0
  Aspartate Aminotransferase: Below | 0 | 0
  Aspartate Aminotransferase: Within | 69 | 42
  Aspartate Aminotransferase: Above | 4 | 3
  Basophils: Unknown | 1 | 0
  Basophils: Below | 0 | 0
  Basophils: Within | 72 | 45
  Basophils: Above | 0 | 0
  Total Bilirubin: Unknown | 0 | 0
  Total Bilirubin: Below | 0 | 0
  Total Bilirubin: Within | 65 | 42
  Total Bilirubin: Above | 8 | 3
  Bilirubin Conjugated/Direct: Unknown | 0 | 0
  Bilirubin Conjugated/Direct: Below | 0 | 0
  Bilirubin Conjugated/Direct: Within | 73 | 44
  Bilirubin Conjugated/Direct: Above | 0 | 1
  Creatinine: Unknown | 0 | 0
  Creatinine: Below | 4 | 7
  Creatinine: Within | 66 | 38
  Creatinine: Above | 3 | 0
  Eosinophils: Unknown | 1 | 0
  Eosinophils: Below | 13 | 6
  Eosinophils: Within | 57 | 39
  Eosinophils: Above | 2 | 0
  Glucose: Unknown | 0 | 0
  Glucose: Below | 2 | 1
  Glucose: Within | 62 | 34
  Glucose: Above | 9 | 10
  Bicarbonate: Unknown | 0 | 0
  Bicarbonate: Below | 7 | 1
  Bicarbonate: Within | 66 | 44
  Bicarbonate: Above | 0 | 0
  Haemoglobin: Unknown | 1 | 0
  Haemoglobin: Below | 12 | 3
  Haemoglobin: Within | 57 | 40
  Haemoglobin: Above | 3 | 2
  Potassium: Unknown | 0 | 0
  Potassium: Below | 0 | 1
  Potassium: Within | 73 | 44
  Potassium: Above | 0 | 0
  Lymphocytes: Unknown | 1 | 0
  Lymphocytes: Below | 1 | 0
  Lymphocytes: Within | 71 | 45
  Lymphocytes: Above | 0 | 0
  Monocytes: Unknown | 1 | 0
  Monocytes: Below | 6 | 3
  Monocytes: Within | 66 | 42
  Monocytes: Above | 0 | 0
  Sodium: Unknown | 0 | 0
  Sodium: Below | 0 | 1
  Sodium: Within | 73 | 44
  Sodium: Above | 0 | 0
  Neutrophils: Unknown | 1 | 0
  Neutrophils: Below | 8 | 3
  Neutrophils: Within | 64 | 40
  Neutrophils: Above | 0 | 2
  Platelets: Unknown | 1 | 0
  Platelets: Below | 2 | 3
  Platelets: Within | 70 | 42
  Platelets: Above | 0 | 0
  White Blood Cells: Unknown | 1 | 0
  White Blood Cells: Below | 5 | 4
  White Blood Cells: Within | 67 | 39
  White Blood Cells: Above | 0 | 2

10. Primary Outcome: Number of Subjects With Any Hematological and Biochemical Parameters Below, Within or Above Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 71 | 47
Participants
  Alanine Aminotransferase: Unknown | 0 | 1
  Alanine Aminotransferase: Below | 0 | 0
  Alanine Aminotransferase: Within | 67 | 40
  Alanine Aminotransferase: Above | 4 | 6
  Albumin: Unknown | 0 | 1
  Albumin: Below | 0 | 0
  Albumin: Within | 67 | 44
  Albumin: Above | 4 | 2
  Alkaline Phosphatase: Unknown | 0 | 1
  Alkaline Phosphatase: Below | 0 | 0
  Alkaline Phosphatase: Within | 68 | 42
  Alkaline Phosphatase: Above | 3 | 4
  Aspartate Aminotransferase: Unknown | 0 | 1
  Aspartate Aminotransferase: Below | 0 | 0
  Aspartate Aminotransferase: Within | 67 | 43
  Aspartate Aminotransferase: Above | 4 | 3
  Basophils: Unknown | 1 | 2
  Basophils: Below | 0 | 0
  Basophils: Within | 70 | 45
  Basophils: Above | 0 | 0
  Total Bilirubin: Unknown | 0 | 1
  Total Bilirubin: Below | 0 | 0
  Total Bilirubin: Within | 64 | 44
  Total Bilirubin: Above | 7 | 2
  Bilirubin Conjugated/Direct: Unknown | 0 | 1
  Bilirubin Conjugated/Direct: Below | 0 | 0
  Bilirubin Conjugated/Direct: Within | 69 | 46
  Bilirubin Conjugated/Direct: Above | 2 | 0
  Creatinine: Unknown | 0 | 1
  Creatinine: Below | 5 | 7
  Creatinine: Within | 65 | 39
  Creatinine: Above | 1 | 0
  Eosinophils: Unknown | 1 | 2
  Eosinophils: Below | 9 | 7
  Eosinophils: Within | 61 | 37
  Eosinophils: Above | 0 | 1
  Glucose: Unknown | 0 | 1
  Glucose: Below | 2 | 0
  Glucose: Within | 59 | 38
  Glucose: Above | 10 | 8
  Bicarbonate: Unknown | 0 | 1
  Bicarbonate: Below | 2 | 0
  Bicarbonate: Within | 69 | 46
  Bicarbonate: Above | 0 | 0
  Haemoglobin: Unknown | 1 | 2
  Haemoglobin: Below | 15 | 5
  Haemoglobin: Within | 53 | 38
  Haemoglobin: Above | 2 | 2
  Potassium: Unknown | 0 | 1
  Potassium: Below | 0 | 0
  Potassium: Within | 70 | 46
  Potassium: Above | 1 | 0
  Lymphocytes: Unknown | 1 | 2
  Lymphocytes: Below | 0 | 1
  Lymphocytes: Within | 68 | 44
  Lymphocytes: Above | 2 | 0
  Monocytes: Unknown | 1 | 2
  Monocytes: Below | 4 | 4
  Monocytes: Within | 66 | 41
  Monocytes: Above | 0 | 0
  Sodium: Unknown | 0 | 1
  Sodium: Below | 0 | 0
  Sodium: Within | 70 | 46
  Sodium: Above | 1 | 0
  Neutrophils: Unknown | 1 | 2
  Neutrophils: Below | 7 | 1
  Neutrophils: Within | 63 | 43
  Neutrophils: Above | 0 | 1
  Platelets: Unknown | 1 | 2
  Platelets: Below | 1 | 2
  Platelets: Within | 69 | 43
  Platelets: Above | 0 | 0
  White Blood Cells: Unknown | 1 | 2
  White Blood Cells: Below | 6 | 2
  White Blood Cells: Within | 64 | 41
  White Blood Cells: Above | 0 | 2

11. Primary Outcome: Number of Subjects With Any Hematological and Biochemical Parameters Below, Within or Above Normal Laboratory Ranges
Description: The assessed parameters were Alanine Aminotransferase, Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Basophils, Bilirubin Total, Bilirubin Conjugated / Direct, Creatinine, Eosinophils, Glucose, Bicarbonate, Haemoglobin, Potassium, Lymphocytes, Monocytes, Sodium, Neutrophils, Platelets and White Blood Cells. Tabulation was made by relation to the normal laboratory ranges: below, within or above, and also staus unknown.
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 72 | 47
Participants
  Alanine Aminotransferase: Unknown | 1 | 2
  Alanine Aminotransferase: Below | 0 | 0
  Alanine Aminotransferase: Within | 66 | 36
  Alanine Aminotransferase: Above | 5 | 9
  Albumin: Unknown | 1 | 2
  Albumin: Below | 0 | 0
  Albumin: Within | 67 | 43
  Albumin: Above | 4 | 2
  Alkaline Phosphatase: Unknown | 1 | 2
  Alkaline Phosphatase: Below | 0 | 0
  Alkaline Phosphatase: Within | 67 | 40
  Alkaline Phosphatase: Above | 4 | 5
  Aspartate Aminotransferase: Unknown | 1 | 2
  Aspartate Aminotransferase: Below | 0 | 0
  Aspartate Aminotransferase: Within | 68 | 41
  Aspartate Aminotransferase: Above | 3 | 4
  Basophils: Unknown | 0 | 1
  Basophils: Below | 0 | 0
  Basophils: Within | 72 | 46
  Basophils: Above | 0 | 0
  Total Bilirubin: Unknown | 1 | 2
  Total Bilirubin: Below | 0 | 0
  Total Bilirubin: Within | 61 | 43
  Total Bilirubin: Above | 10 | 2
  Bilirubin Conjugated/Direct: Unknown | 1 | 2
  Bilirubin Conjugated/Direct: Below | 0 | 0
  Bilirubin Conjugated/Direct: Within | 70 | 44
  Bilirubin Conjugated/Direct: Above | 1 | 1
  Creatinine: Unknown | 1 | 2
  Creatinine: Below | 5 | 7
  Creatinine: Within | 66 | 37
  Creatinine: Above | 0 | 1
  Eosinophils: Unknown | 0 | 1
  Eosinophils: Below | 12 | 5
  Eosinophils: Within | 59 | 41
  Eosinophils: Above | 1 | 0
  Glucose: Unknown | 1 | 2
  Glucose: Below | 2 | 0
  Glucose: Within | 62 | 38
  Glucose: Above | 7 | 7
  Bicarbonate: Unknown | 1 | 2
  Bicarbonate: Below | 5 | 2
  Bicarbonate: Within | 66 | 43
  Bicarbonate: Above | 0 | 0
  Haemoglobin: Unknown | 0 | 1
  Haemoglobin: Below | 14 | 5
  Haemoglobin: Within | 57 | 37
  Haemoglobin: Above | 1 | 4
  Potassium: Unknown | 1 | 2
  Potassium: Below | 0 | 0
  Potassium: Within | 71 | 45
  Potassium: Above | 0 | 0
  Lymphocytes: Unknown | 0 | 1
  Lymphocytes: Below | 0 | 0
  Lymphocytes: Within | 72 | 46
  Lymphocytes: Above | 0 | 0
  Monocytes: Unknown | 0 | 1
  Monocytes: Below | 6 | 6
  Monocytes: Within | 66 | 40
  Monocytes: Above | 0 | 0
  Sodium: Unknown | 1 | 2
  Sodium: Below | 0 | 0
  Sodium: Within | 71 | 45
  Sodium: Above | 0 | 0
  Neutrophils: Unknown | 0 | 1
  Neutrophils: Below | 6 | 5
  Neutrophils: Within | 66 | 39
  Neutrophils: Above | 0 | 2
  Platelets: Unknown | 0 | 1
  Platelets: Below | 3 | 2
  Platelets: Within | 69 | 44
  Platelets: Above | 0 | 0
  White Blood Cells: Unknown | 0 | 1
  White Blood Cells: Below | 5 | 7
  White Blood Cells: Within | 67 | 37
  White Blood Cells: Above | 0 | 2

12. Primary Outcome: Number of Subjects With Any Hematological and Biochemical Parameters Below, Within or Above Normal Laboratory Ranges
Description: as for outcome 8
Time Frame: At Month 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 71 | 47
Participants
  Alanine Aminotransferase: Unknown | 0 | 0
  Alanine Aminotransferase: Below | 0 | 0
  Alanine Aminotransferase: Within | 67 | 41
  Alanine Aminotransferase: Above | 4 | 6
  Albumin: Unknown | 0 | 0
  Albumin: Below | 0 | 0
  Albumin: Within | 68 | 44
  Albumin: Above | 3 | 3
  Alkaline Phosphatase: Unknown | 0 | 0
  Alkaline Phosphatase: Below | 0 | 0
  Alkaline Phosphatase: Within | 67 | 42
  Alkaline Phosphatase: Above | 4 | 5
  Aspartate Aminotransferase: Unknown | 0 | 0
  Aspartate Aminotransferase: Below | 0 | 0
  Aspartate Aminotransferase: Within | 66 | 45
  Aspartate Aminotransferase: Above | 5 | 2
  Basophils: Unknown | 2 | 1
  Basophils: Below | 0 | 0
  Basophils: Within | 69 | 46
  Basophils: Above | 0 | 0
  Total Bilirubin: Unknown | 0 | 0
  Total Bilirubin: Below | 0 | 0
  Total Bilirubin: Within | 60 | 45
  Total Bilirubin: Above | 11 | 2
  Bilirubin Conjugated/Direct: Unknown | 0 | 0
  Bilirubin Conjugated/Direct: Below | 0 | 0
  Bilirubin Conjugated/Direct: Within | 68 | 46
  Bilirubin Conjugated/Direct: Above | 3 | 1
  Creatinine: Unknown | 0 | 0
  Creatinine: Below | 7 | 7
  Creatinine: Within | 62 | 39
  Creatinine: Above | 2 | 1
  Eosinophils: Unknown | 2 | 1
  Eosinophils: Below | 13 | 9
  Eosinophils: Within | 55 | 36
  Eosinophils: Above | 1 | 1
  Glucose: Unknown | 0 | 0
  Glucose: Below | 1 | 1
  Glucose: Within | 62 | 37
  Glucose: Above | 8 | 9
  Bicarbonate: Unknown | 0 | 0
  Bicarbonate: Below | 7 | 7
  Bicarbonate: Within | 63 | 40
  Bicarbonate: Above | 1 | 0
  Haemoglobin: Unknown | 2 | 1
  Haemoglobin: Below | 13 | 6
  Haemoglobin: Within | 55 | 37
  Haemoglobin: Above | 1 | 3
  Potassium: number analyzed (Participants) | 70 | 47
  Potassium: Unknown | 0 | 0
  Potassium: Below | 0 | 0
  Potassium: Within | 70 | 47
  Potassium: Above | 0 | 0
  Lymphocytes: Unknown | 2 | 1
  Lymphocytes: Below | 4 | 3
  Lymphocytes: Within | 65 | 42
  Lymphocytes: Above | 0 | 1
  Monocytes: Unknown | 2 | 1
  Monocytes: Below | 2 | 4
  Monocytes: Within | 67 | 42
  Monocytes: Above | 0 | 0
  Sodium: Unknown | 0 | 0
  Sodium: Below | 0 | 0
  Sodium: Within | 71 | 47
  Sodium: Above | 0 | 0
  Neutrophils: Unknown | 2 | 1
  Neutrophils: Below | 5 | 5
  Neutrophils: Within | 64 | 37
  Neutrophils: Above | 0 | 4
  Platelets: Unknown | 2 | 1
  Platelets: Below | 2 | 2
  Platelets: Within | 67 | 44
  Platelets: Above | 0 | 0
  White Blood Cells: Unknown | 2 | 1
  White Blood Cells: Below | 6 | 4
  White Blood Cells: Within | 62 | 39
  White Blood Cells: Above | 1 | 3

13. Primary Outcome: Number of Subjects With Any Hematological and Biochemical Parameters Below, Within or Above Normal Laboratory Ranges
Description: as for outcome 11
Time Frame: At Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 68 | 47
Participants
  Alanine Aminotransferase: Unknown | 1 | 1
  Alanine Aminotransferase: Below | 0 | 0
  Alanine Aminotransferase: Within | 64 | 42
  Alanine Aminotransferase: Above | 3 | 4
  Albumin: Unknown | 1 | 1
  Albumin: Below | 0 | 1
  Albumin: Within | 64 | 41
  Albumin: Above | 3 | 4
  Alkaline Phosphatase: Unknown | 1 | 1
  Alkaline Phosphatase: Below | 0 | 0
  Alkaline Phosphatase: Within | 63 | 42
  Alkaline Phosphatase: Above | 4 | 4
  Aspartate Aminotransferase: Unknown | 1 | 1
  Aspartate Aminotransferase: Below | 0 | 0
  Aspartate Aminotransferase: Within | 65 | 43
  Aspartate Aminotransferase: Above | 2 | 3
  Basophils: Unknown | 0 | 0
  Basophils: Below | 0 | 0
  Basophils: Within | 68 | 47
  Basophils: Above | 0 | 0
  Total Bilirubin: Unknown | 1 | 1
  Total Bilirubin: Below | 0 | 0
  Total Bilirubin: Within | 57 | 43
  Total Bilirubin: Above | 10 | 3
  Bilirubin Conjugated/Direct: Unknown | 1 | 1
  Bilirubin Conjugated/Direct: Below | 0 | 0
  Bilirubin Conjugated/Direct: Within | 67 | 46
  Bilirubin Conjugated/Direct: Above | 0 | 0
  Creatinine: Unknown | 1 | 1
  Creatinine: Below | 7 | 6
  Creatinine: Within | 57 | 39
  Creatinine: Above | 3 | 1
  Eosinophils: Unknown | 0 | 0
  Eosinophils: Below | 11 | 7
  Eosinophils: Within | 56 | 39
  Eosinophils: Above | 1 | 1
  Glucose: Unknown | 1 | 1
  Glucose: Below | 0 | 0
  Glucose: Within | 63 | 39
  Glucose: Above | 4 | 7
  Bicarbonate: Unknown | 1 | 1
  Bicarbonate: Below | 6 | 4
  Bicarbonate: Within | 61 | 42
  Bicarbonate: Above | 0 | 0
  Haemoglobin: Unknown | 0 | 0
  Haemoglobin: Below | 19 | 6
  Haemoglobin: Within | 49 | 40
  Haemoglobin: Above | 0 | 1
  Potassium: Unknown | 1 | 1
  Potassium: Below | 1 | 0
  Potassium: Within | 66 | 46
  Potassium: Above | 0 | 0
  Lymphocytes: Unknown | 0 | 0
  Lymphocytes: Below | 0 | 1
  Lymphocytes: Within | 67 | 46
  Lymphocytes: Above | 1 | 0
  Monocytes: Unknown | 0 | 0
  Monocytes: Below | 5 | 2
  Monocytes: Within | 63 | 45
  Monocytes: Above | 0 | 0
  Sodium: Unknown | 1 | 1
  Sodium: Below | 0 | 0
  Sodium: Within | 67 | 46
  Sodium: Above | 0 | 0
  Neutrophils: Unknown | 0 | 0
  Neutrophils: Below | 7 | 1
  Neutrophils: Within | 61 | 44
  Neutrophils: Above | 0 | 2
  Platelets: Unknown | 0 | 0
  Platelets: Below | 2 | 1
  Platelets: Within | 66 | 46
  Platelets: Above | 0 | 0
  White Blood Cells: Unknown | 0 | 0
  White Blood Cells: Below | 6 | 1
  White Blood Cells: Within | 62 | 44
  White Blood Cells: Above | 0 | 2

14. Primary Outcome: Number of Subjects With Any Significant Change in Antiretroviral Therapy (ART), Including Initiation of ART in ART-naïve Subjects
Description: In this analysis, results were tabulated for the main study groups. Significant changes to ART appeared due to failure to control HIV viral load and due to failure to maintain high CD4 cells count.
Time Frame: From Month 0 until Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants
  Failure to control HIV viral load | 0 | 0
  Failure to maintain high CD4 cells count | 0 | 0

15. Primary Outcome: Number of Subjects With Any AIDS-defining Condition
Description: In this analysis, results were tabulated for the main study groups.
Time Frame: From Month 0 until Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants | 0 | 0

16. Primary Outcome: Number of Subjects With Any Pre-defined Changes in HIV Viral Load (VL) and CD4 T-cell Count
Description: In this analysis, results were tabulated for the main study groups.
Time Frame: From Month 1 to Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants
  Change in HIV viral load | 3 | 1
  Change in CD4 cells count | 7 | 4

17. Primary Outcome: Number of Subjects With Any Significant Change in Antiretroviral Therapy (ART), Including Initiation of ART in ART-naïve Subjects, by HIV Status
Description: In this analysis, results were tabulated by HIV status
Time Frame: From Month 0 to Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A: ART-treated subjects with a high CD4 T-cells count: ≥ 200 cells/mm3, receiving three doses of GSK 1437173A vaccine (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
- ART High CD4 Cohort - Placebo; ART Low CD4 Cohort - Placebo; Non-ART High CD4 Cohort - Placebo: ART-naïve HIV-infected subjects with a high CD4 T-cells count of ≥ 500 cells/mm3, receiving three doses of placebo (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
- ART Low CD4 Cohort - GSK 1437173A: ART-treated subjects with a low CD4 T-cells count: 50-199 cells/mm3, receiving three doses of GSK 1437173A vaccine (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
- Non-ART High CD4 Cohort - GSK 1437173A: ART-naïve HIV-infected subjects with a high CD4 T-cells count of ≥ 500 cells/mm3, receiving three doses of GSK 1437173A vaccine (Months 0, 2 and 6), administered intramuscularly, in the deltoid muscle of the non-dominant arm.
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 56 | 38 | 9 | 5 | 9 | 6
Participants
  Due to failure to control HIV viral load | 0 | 0 | 0 | 0 | 0 | 0
  Due to failure to maintain high CD4 cells count | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Subjects With Any AIDS-defining Condition, by HIV Status
Description: In this analysis, results were tabulated by HIV status
Time Frame: From Month 0 to Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 56 | 38 | 9 | 5 | 9 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Number of Subjects With Any Pre-defined Changes in HIV Viral Load (VL) and CD4 T-cell Count, by HIV Status
Description: In this analysis, results were tabulated by HIV status.
Time Frame: From Month 1 to Month 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 56 | 38 | 9 | 5 | 9 | 6
Participants
  Change in HIV viral load | 1 | 0 | 1 | 0 | 1 | 1
  Change in CD4 cells count | 5 | 3 | 1 | 1 | 1 | 0

20. Primary Outcome: Frequency of gE-specific CD4 T-cells
Description: The analysis focused on CD4 T-cells expressing at least 2 cytokines (among interferon-gamma (IFN-g) , interleukin-2 (IL-2), tumour necrosis factor-alpha (TNF-a) and/or CD40 ligand (CD40L)) as determined by in vitro intracellular cytokine staining (ICS) at Month 7 in ART and non-ART cohorts presenting high CD4 counts at enrollment.
Time Frame: At Month 7
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available at Month 7.
Measure: Mean (Standard Deviation); unit: CD4 T-cells/million T-cells
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 30 | 20
CD4 T-cells/million T-cells | 4684.50 (5376.83) | 158.64 (151.15)

21. Primary Outcome: -Anti-gE Antibody (Ab) Concentrations
Description: -Anti-gE antibody (Ab) concentrations were determined by Enzyme-Linked Immunosorbent Assay (ELISA) at Month 7 in ART and non-ART cohorts presenting high CD4 counts at enrolment. Antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in milli-international units per milliliter (mIU/mL).
Time Frame: At Month 7
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 54 | 36
mIU/mL | 63812.6 [51183.6 to 79557.7] | 1028.4 [658.9 to 1605.0]

22. Secondary Outcome: -Frequencies of Varicella-Zoster Virus (VZV)- and gE-specific CD4 T-cells
Description: The analysis focused on CD4 T cells expressing at least 2 cytokines (among IFN-g, IL-2, TNF-a and/or CD40L as determined by ICS at Months 0, 1, 2, 3, 6, 7 and 18 and tabulated for the main study groups.
Time Frame: At Month 0, 1, 2, 3, 6, 7 and 18
Population: The analysis was performed on the ATP cohorts for immunogenicity and for persistence, which included all evaluable subjects for whom data concerning immunogenicity measures were available at the considered time points (up to Month 7 for the ATP cohort for immunogenicity and at Month 18 for the ATP cohort for persistence).
Measure: Mean (Standard Deviation); unit: CD4 T-cells/million T-cells
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 49 | 35
CD4 T-cells/million T-cells
  VZV-specific CD4 [2+] T-cells, pre-vaccination: number analyzed (Participants) | 32 | 27
  VZV-specific CD4 [2+] T-cells, pre-vaccination | 750.20 (989.36) | 835.80 (1949.39)
  VZV-specific CD4 [2+] T-cells, Month 1: number analyzed (Participants) | 40 | 26
  VZV-specific CD4 [2+] T-cells, Month 1 | 768.60 (739.68) | 913.87 (2262.66)
  VZV-specific CD4 [2+] T-cells, Month 2: number analyzed (Participants) | 37 | 26
  VZV-specific CD4 [2+] T-cells, Month 2 | 734.09 (680.34) | 874.13 (2027.95)
  VZV-specific CD4 [2+] T-cells, Month 3: number analyzed (Participants) | 41 | 28
  VZV-specific CD4 [2+] T-cells, Month 3 | 1878.81 (1615.20) | 987.24 (1988.86)
  VZV-specific CD4 [2+] T-cells, Month 6: number analyzed (Participants) | 29 | 19
  VZV-specific CD4 [2+] T-cells, Month 6 | 1646.83 (1202.32) | 674.20 (657.00)
  VZV-specific CD4 [2+] T-cells, Month 7: number analyzed (Participants) | 30 | 20
  VZV-specific CD4 [2+] T-cells, Month 7 | 2626.71 (2514.40) | 1204.44 (1911.53)
  VZV-specific CD4 [2+] T-cells, Month 18: number analyzed (Participants) | 48 | 35
  VZV-specific CD4 [2+] T-cells, Month 18 | 995.35 (842.96) | 531.24 (579.63)
  gE-specific CD4 [2+] T-cells, pre-vaccination: number analyzed (Participants) | 33 | 27
  gE-specific CD4 [2+] T-cells, pre-vaccination | 218.26 (254.94) | 123.15 (170.79)
  gE-specific CD4 [2+] T-cells, Month 1: number analyzed (Participants) | 40 | 26
  gE-specific CD4 [2+] T-cells, Month 1 | 704.06 (614.49) | 132.49 (213.05)
  gE-specific CD4 [2+] T-cells, Month 2: number analyzed (Participants) | 38 | 26
  gE-specific CD4 [2+] T-cells, Month 2 | 649.68 (555.51) | 140.95 (197.99)
  gE-specific CD4 [2+] T-cells, Month 3: number analyzed (Participants) | 41 | 28
  gE-specific CD4 [2+] T-cells, Month 3 | 3503.69 (2971.74) | 160.10 (220.32)
  gE-specific CD4 [2+] T-cells, Month 6: number analyzed (Participants) | 29 | 19
  gE-specific CD4 [2+] T-cells, Month 6 | 2647.71 (1972.00) | 133.70 (137.94)
  gE-specific CD4 [2+] T-cells, Month 7: number analyzed (Participants) | 30 | 20
  gE-specific CD4 [2+] T-cells, Month 7 | 4684.50 (5376.83) | 158.64 (151.15)
  gE-specific CD4 [2+] T-cells, Month 18 | 1929.30 (1603.50) | 139.50 (219.57)

23. Secondary Outcome: -Frequencies of Varicella-Zoster Virus (VZV)- and gE-specific CD4 T-cells, by HIV Status
Description: The analysis focused on CD4 T-cells expressing at least 2 cytokines (among IFN-g, IL-2, TNF-a and/or CD40L as determined by ICS at Months 0, 1, 2, 3, 6, 7 and 18 and tabulated by HIV status.
Time Frame: At Months 0, 1, 2, 3, 6, 7 and 18
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: CD4 T-cells/million T-cells
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 40 | 28 | 5 | 3 | 5 | 4
CD4 T-cells/million T-cells
  VZV-specific CD4 [2+] T-cells, pre-vaccination: number analyzed (Participants) | 27 | 24 | 2 | 1 | 3 | 2
  VZV-specific CD4 [2+] T-cells, pre-vaccination | 789.48 (1037.59) | 927.27 (2053.32) | 1.00 (0.00) | 86.96 (NA) — There were not enough subjects for SD analysis to be computed. | 896.13 (749.70) | 112.66 (157.91)
  VZV-specific CD4 [2+] T-cells, Month 1: number analyzed (Participants) | 30 | 22 | 5 | 2 | 5 | 2
  VZV-specific CD4 [2+] T-cells, Month 1 | 830.78 (775.61) | 1049.73 (2442.95) | 114.79 (114.03) | 146.91 (142.99) | 1049.36 (546.09) | 186.38 (31.21)
  VZV-specific CD4 [2+] T-cells, Month 2: number analyzed (Participants) | 28 | 22 | 4 | 2 | 5 | 2
  VZV-specific CD4 [2+] T-cells, Month 2 | 716.33 (699.22) | 991.07 (2190.70) | 814.64 (920.49) | 329.96 (53.46) | 769.13 (469.02) | 131.90 (185.13)
  VZV-specific CD4 [2+] T-cells, Month 3: number analyzed (Participants) | 33 | 22 | 3 | 3 | 5 | 3
  VZV-specific CD4 [2+] T-cells, Month 3 | 1973.47 (1669.57) | 1075.62 (2186.45) | 1804.94 (2350.96) | 408.18 (330.78) | 1298.35 (725.44) | 918.17 (1580.86)
  VZV-specific CD4 [2+] T-cells, Month 6: number analyzed (Participants) | 25 | 16 | 3 | 1 | 1 | 2
  VZV-specific CD4 [2+] T-cells, Month 6 | 1624.32 (1161.05) | 786.72 (657.24) | 1996.37 (1937.58) | 136.42 (NA) — There were not enough subjects for SD analysis to be computed. | 1160.93 (NA) — There were not enough subjects for SD analysis to be computed. | 42.92 (37.09)
  VZV-specific CD4 [2+] T-cells, Month 7: number analyzed (Participants) | 26 | 19 | 3 | 1 | 1 | 0
  VZV-specific CD4 [2+] T-cells, Month 7 | 2285.90 (1998.16) | 1261.84 (1946.12) | 6235.67 (4334.14) | 113.88 (NA) — There were not enough subjects for SD analysis to be computed. | 660.88 (NA) — There were not enough subjects for SD analysis to be computed. |
  VZV-specific CD4 [2+] T-cells, Month 18: number analyzed (Participants) | 40 | 28 | 3 | 3 | 5 | 4
  VZV-specific CD4 [2+] T-cells, Month 18 | 1051.12 (816.86) | 599.00 (587.08) | 853.05 (1235.35) | 580.71 (683.08) | 634.55 (933.54) | 19.77 (22.14)
  gE-specific CD4 [2+] T-cells, pre-vaccination: number analyzed (Participants) | 28 | 24 | 2 | 1 | 3 | 2
  gE-specific CD4 [2+] T-cells, pre-vaccination | 215.99 (266.22) | 136.29 (176.85) | 51.15 (70.92) | 1.00 (NA) — There were not enough subjects for SD analysis to be computed. | 350.86 (161.96) | 26.57 (36.17)
  gE-specific CD4 [2+] T-cells, Month 1: number analyzed (Participants) | 30 | 22 | 5 | 2 | 5 | 2
  gE-specific CD4 [2+] T-cells, Month 1 | 682.62 (595.89) | 134.21 (224.96) | 584.10 (652.67) | 161.73 (227.30) | 952.65 (763.24) | 84.33 (117.84)
  gE-specific CD4 [2+] T-cells, Month 2: number analyzed (Participants) | 29 | 22 | 4 | 2 | 5 | 2
  gE-specific CD4 [2+] T-cells, Month 2 | 610.30 (558.27) | 157.92 (208.48) | 960.39 (632.86) | 94.19 (131.79) | 629.54 (513.99) | 1.00 (0.00)
  gE-specific CD4 [2+] T-cells, Month 3: number analyzed (Participants) | 33 | 22 | 3 | 3 | 5 | 3
  gE-specific CD4 [2+] T-cells, Month 3 | 3722.21 (2789.70) | 190.58 (233.81) | 4754.94 (6004.05) | 1.00 (0.00) | 1310.76 (670.56) | 95.71 (164.04)
  gE-specific CD4 [2+] T-cells, Month 6: number analyzed (Participants) | 25 | 16 | 3 | 1 | 1 | 2
  gE-specific CD4 [2+] T-cells, Month 6 | 2386.40 (1571.28) | 152.52 (141.50) | 5403.79 (3326.03) | 97.99 (NA) — There were not enough subjects for SD analysis to be computed. | 912.30 (NA) — There were not enough subjects for SD analysis to be computed. | 1.00 (0.00)
  gE-specific CD4 [2+] T-cells, Month 7: number analyzed (Participants) | 26 | 19 | 3 | 1 | 1 | 0
  gE-specific CD4 [2+] T-cells, Month 7 | 3649.92 (3112.69) | 166.94 (150.54) | 14925.30 (10934.07) | 1.00 (NA) — There were not enough subjects for SD analysis to be computed. | 861.21 (NA) — There were not enough subjects for SD analysis to be computed. |
  gE-specific CD4 [2+] T-cells, Month 18: number analyzed (Participants) | 40 | 28 | 4 | 3 | 5 | 4
  gE-specific CD4 [2+] T-cells, Month 18 | 2071.17 (1583.58) | 159.05 (239.50) | 2035.18 (2100.82) | 109.97 (93.90) | 709.62 (1011.03) | 24.81 (47.63)

24. Secondary Outcome: -Anti-VZV and Anti-gE Antibody Concentrations
Description: Antibody concentrations were as determined by ELISA and tabulated for the main study groups. Anti-VZV and anti-gE antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in mIU/mL.
Time Frame: At Months 0, 1, 2, 3, 6, 7 and 18
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 54 | 37
mIU/mL
  Anti-VZV, Pre-vaccination: number analyzed (Participants) | 48 | 36
  Anti-VZV, Pre-vaccination | 1292.7 [999.8 to 1671.4] | 1074.7 [672.7 to 1717.0]
  Anti-VZV, Month 1: number analyzed (Participants) | 43 | 33
  Anti-VZV, Month 1 | 6953.8 [5425.1 to 8913.3] | 1173.8 [762.9 to 1805.8]
  Anti-VZV, Month 2: number analyzed (Participants) | 45 | 33
  Anti-VZV, Month 2 | 5170.9 [4032.7 to 6630.4] | 987.6 [596.3 to 1635.8]
  Anti-VZV, Month 3: number analyzed (Participants) | 50 | 33
  Anti-VZV, Month 3 | 11119.7 [9190.8 to 13453.3] | 1037.8 [620.2 to 1736.5]
  Anti-VZV, Month 6: number analyzed (Participants) | 49 | 34
  Anti-VZV, Month 6 | 8244.0 [6678.6 to 10176.3] | 1069.8 [653.3 to 1751.7]
  Anti-VZV, Month 7: number analyzed (Participants) | 49 | 32
  Anti-VZV, Month 7 | 14560.8 [11849.0 to 17893.1] | 999.3 [598.3 to 1669.2]
  Anti-VZV, Month 18: number analyzed (Participants) | 46 | 29
  Anti-VZV, Month 18 | 7493.3 [5926.7 to 9473.9] | 922.9 [521.1 to 1634.6]
  Anti-gE, Pre-vaccination: number analyzed (Participants) | 53 | 37
  Anti-gE, Pre-vaccination | 1218.4 [895.0 to 1658.7] | 849.5 [551.1 to 1309.4]
  Anti-gE, Month 1: number analyzed (Participants) | 54 | 36
  Anti-gE, Month 1 | 24113.2 [18317.4 to 31743.0] | 1059.0 [749.4 to 1496.5]
  Anti-gE, Month 2: number analyzed (Participants) | 53 | 37
  Anti-gE, Month 2 | 17112.6 [12929.5 to 22649.1] | 903.3 [590.9 to 1380.9]
  Anti-gE, Month 3 | 50443.0 [40899.6 to 62213.2] | 992.9 [647.4 to 1522.6]
  Anti-gE, Month 6 | 34159.4 [27221.0 to 42866.2] | 1013.1 [660.5 to 1553.7]
  Anti-gE, Month 7 | 63812.6 [51183.6 to 79557.7] | 1028.4 [658.9 to 1605.0]
  Anti-gE, Month 18: number analyzed (Participants) | 49 | 37
  Anti-gE, Month 18 | 25242.2 [19618.9 to 32477.3] | 918.0 [588.0 to 1433.1]

25. Secondary Outcome: -Anti-VZV and Anti-gE Antibody Concentrations, by HIV Status
Description: Antibody concentrations were as determined by ELISA and tabulated by HIV status. Anti-VZV and anti-gE antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in mIU/mL.
Time Frame: At Months 0, 1, 2, 3, 6, 7 and 18
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 44 | 30 | 5 | 4 | 5 | 4
mIU/mL
  Anti-VZV, Pre-vaccination: number analyzed (Participants) | 38 | 29 | 5 | 3 | 5 | 4
  Anti-VZV, Pre-vaccination | 1161.5 [900.3 to 1498.6] | 985.1 [568.7 to 1706.4] | 2272.6 [559.1 to 9236.6] | 2511.9 [693.0 to 9104.4] | 1658.0 [315.9 to 8701.1] | 1068.5 [117.3 to 9735.4]
  Anti-VZV, Month 1: number analyzed (Participants) | 34 | 26 | 4 | 3 | 5 | 4
  Anti-VZV, Month 1 | 7017.8 [5441.2 to 9051.3] | 1059.6 [641.1 to 1751.2] | 6731.0 [572.7 to 79107.0] | 2871.0 [1386.7 to 5944.3] | 6706.0 [2477.9 to 18148.5] | 1167.3 [130.1 to 10475.4]
  Anti-VZV, Month 2: number analyzed (Participants) | 38 | 27 | 4 | 2 | 3 | 4
  Anti-VZV, Month 2 | 5056.5 [3973.9 to 6434.0] | 886.9 [498.6 to 1577.4] | 5649.6 [418.4 to 76276.9] | 2902.1 [1.9 to 4493973] | 6100.0 [480.4 to 77462.7] | 1191.1 [119.6 to 11860.7]
  Anti-VZV, Month 3: number analyzed (Participants) | 41 | 28 | 5 | 1 | 4 | 4
  Anti-VZV, Month 3 | 11631.9 [9523.8 to 14206.6] | 1002.7 [565.8 to 1777.1] | 9110.7 [2224.8 to 37308.9] | 2479.3 [NA to NA] — There were not enough subjects for a Lower Limit (LL) and Upper Limit (UL) to be computed. | 8990.7 [5233.1 to 15446.6] | 1062.0 [81.1 to 13906.2]
  Anti-VZV, Month 6: number analyzed (Participants) | 39 | 27 | 5 | 3 | 5 | 4
  Anti-VZV, Month 6 | 9027.6 [7225.1 to 11279.6] | 957.0 [537.2 to 1705.0] | 7634.7 [2054.6 to 28369.5] | 3164.8 [510.5 to 19621.7] | 4384.3 [2322.5 to 8276.5] | 1006.3 [115.7 to 8754.6]
  Anti-VZV, Month 7: number analyzed (Participants) | 40 | 26 | 5 | 2 | 4 | 4
  Anti-VZV, Month 7 | 15278.5 [12420.2 to 18794.5] | 930.5 [511.6 to 1692.3] | 14763.2 [2859.6 to 76216.1] | 2177.3 [8.7 to 544573.1] | 8845.8 [5463.6 to 14321.5] | 1076.7 [109.5 to 10591.1]
  Anti-VZV, Month 18: number analyzed (Participants) | 37 | 24 | 4 | 2 | 5 | 3
  Anti-VZV, Month 18 | 8242.2 [6484.1 to 10476.9] | 838.1 [435.9 to 1611.5] | 6106.2 [748.6 to 49809.5] | 1955.3 [188.8 to 20249.5] | 4361.7 [1721.5 to 11050.9] | 1209.2 [13.9 to 105230.8]
  Anti-gE, Pre-vaccination: number analyzed (Participants) | 43 | 30 | 5 | 3 | 5 | 4
  Anti-gE, Pre-vaccination | 1113.2 [794.3 to 1560.3] | 791.0 [490.7 to 1275.1] | 1845.1 [465.1 to 7319.1] | 2420.7 [512.0 to 11445.2] | 1748.6 [308.5 to 9912.2] | 661.2 [43.8 to 9984.8]
  Anti-gE, Month 1: number analyzed (Participants) | 44 | 29 | 5 | 3 | 5 | 4
  Anti-gE, Month 1 | 25530.6 [19158.6 to 34021.9] | 1029.5 [719.5 to 1473.1] | 18767.2 [2219.4 to 158697.1] | 2328.1 [446.4 to 12141.8] | 18742.3 [6616.7 to 53089.1] | 720.0 [50.6 to 10238.5]
  Anti-gE, Month 2: number analyzed (Participants) | 43 | 30 | 5 | 3 | 5 | 4
  Anti-gE, Month 2 | 18208.6 [13537.4 to 24491.6] | 839.8 [524.6 to 1344.4] | 13106.4 [1619.0 to 106104.2] | 2465.5 [561.9 to 10817.4] | 13100.6 [4828.6 to 35543.7] | 735.0 [52.7 to 10245.9]
  Anti-gE, Month 3: number analyzed (Participants) | 44 | 30 | 5 | 3 | 5 | 4
  Anti-gE, Month 3 | 54777.7 [44077.1 to 68076.1] | 955.6 [590.6 to 1546.2] | 36592.6 [7026.0 to 190581.1] | 2166.3 [618.9 to 7583.1] | 33662.4 [20665.6 to 54833.0] | 736.6 [52.1 to 10414.5]
  Anti-gE, Month 6: number analyzed (Participants) | 44 | 30 | 5 | 3 | 5 | 4
  Anti-gE, Month 6 | 38068.2 [29964.3 to 48363.7] | 932.8 [582.6 to 1493.3] | 24725.0 [5143.2 to 118862.3] | 2629.2 [561.7 to 12306.8] | 18189.6 [11258.0 to 29389.0] | 920.6 [54.8 to 15461.5]
  Anti-gE, Month 7: number analyzed (Participants) | 44 | 29 | 5 | 3 | 5 | 4
  Anti-gE, Month 7 | 71309.6 [57019.3 to 89181.5] | 928.8 [566.8 to 1522.1] | 47382.6 [9151.2 to 245336.2] | 2553.0 [610.1 to 10683.1] | 32334.6 [17277.6 to 60513.4] | 1087.6 [60.2 to 19641.4]
  Anti-gE, Month 18: number analyzed (Participants) | 40 | 29 | 4 | 4 | 5 | 4
  Anti-gE, Month 18 | 28854.6 [22512.5 to 36983.3] | 849.4 [514.6 to 1401.9] | 18995.8 [1733.3 to 208181.4] | 1953.7 [572.7 to 6665.3] | 10869.2 [4435.4 to 26635.7] | 757.8 [34.8 to 16519.1]

26. Secondary Outcome: Number of Subjects With Any Herpes Zoster (HZ) Cases and Complications
Time Frame: From Month 0 until Month 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1437173A Group | Placebo Group
Number analyzed (Participants) | 74 | 49
Participants | 1 | 0

27. Secondary Outcome: CD4 Count
Description: CD4 count was tabulated by HIV status.
Time Frame: At Screening Visit (up to 21 days prior to Month 0), Months 1, 2, 3, 6, 7 and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CD4 T-cells/million T-cells
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 56 | 38 | 9 | 5 | 9 | 6
CD4 T-cells/million T-cells
  CD4+, pre-vaccination | 631.46 (236.36) | 683.39 (228.29) | 152.11 (38.39) | 132.20 (11.19) | 805.33 (132.38) | 901.67 (177.61)
  CD4+, Month 1: number analyzed (Participants) | 55 | 35 | 9 | 5 | 9 | 5
  CD4+, Month 1 | 630.55 (241.78) | 694.69 (307.98) | 151.11 (38.72) | 163.00 (53.66) | 879.67 (277.37) | 773.40 (144.85)
  CD4+, Month 2: number analyzed (Participants) | 54 | 36 | 8 | 4 | 8 | 5
  CD4+, Month 2 | 667.69 (309.22) | 656.14 (262.43) | 131.13 (39.57) | 133.75 (31.86) | 808.75 (211.32) | 804.00 (199.09)
  CD4+, Month 3: number analyzed (Participants) | 55 | 36 | 9 | 5 | 8 | 5
  CD4+, Month 3 | 633.60 (228.75) | 640.14 (238.05) | 153.11 (54.27) | 142.60 (36.49) | 783.63 (239.92) | 762.60 (185.66)
  CD4+, Month 6: number analyzed (Participants) | 53 | 36 | 9 | 5 | 7 | 5
  CD4+, Month 6 | 655.02 (264.67) | 668.28 (308.64) | 145.33 (29.74) | 145.20 (43.18) | 776.43 (303.30) | 1082.80 (649.82)
  CD4+, Month 7: number analyzed (Participants) | 54 | 37 | 8 | 5 | 7 | 5
  CD4+, Month 7 | 654.69 (271.31) | 658.81 (246.53) | 170.25 (44.52) | 150.40 (35.11) | 869.14 (297.04) | 866.00 (144.30)
  CD4+, Month 18: number analyzed (Participants) | 51 | 35 | 7 | 5 | 7 | 5
  CD4+, Month 18 | 679.71 (247.57) | 651.06 (247.30) | 168.43 (58.49) | 151.40 (57.48) | 720.00 (228.77) | 824.40 (207.57)

28. Secondary Outcome: HIV VL
Description: HIV VL was tabulated by HIV status, for subjects with a number of available results greater than or equal to (≥) 40 copies/mL.
Time Frame: At Screening Visit (up to 21 days prior to Month 0), Months 1, 2, 3, 6, 7 and 18
Population: The analysis was performed on the Total Vaccinated cohort, which included only vaccinated subjects with at least one vaccine administration documented, who had available results of ≥ 40 copies/mL.
Measure: Mean (Standard Deviation); unit: HIV-RNA copies/mL
Arm/Group | Antiretroviral Therapy (ART) High CD4 Cohort - GSK 1437173A | ART High CD4 Cohort - Placebo | ART Low CD4 Cohort - GSK 1437173A | ART Low CD4 Cohort - Placebo | Non-ART High CD4 Cohort - GSK 1437173A | Non-ART High CD4 Cohort - Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 1 | 9 | 6
HIV-RNA copies/mL
  HIV VL, pre-vaccination: number analyzed (Participants) | 0 | 0 | 1 | 0 | 9 | 6
  HIV VL, pre-vaccination |  |  | 62.00 (NA) — There were not enough subjects for SD analysis to be computed. |  | 23014.11 (18435.10) | 16022.17 (23652.18)
  HIV VL, Month 1: number analyzed (Participants) | 1 | 0 | 1 | 0 | 9 | 5
  HIV VL, Month 1 | 42.00 (NA) — There were not enough subjects for SD analysis to be computed. |  | 48.00 (NA) — There were not enough subjects for SD analysis to be computed. |  | 24538.89 (19056.10) | 14415.80 (9289.92)
  HIV VL, Month 2: number analyzed (Participants) | 3 | 1 | 2 | 0 | 8 | 4
  HIV VL, Month 2 | 48.67 (10.79) | 55.00 (NA) — There were not enough subjects for SD analysis to be computed. | 48.00 (2.83) |  | 24134.25 (13753.92) | 18188.25 (15199.35)
  HIV VL, Month 3: number analyzed (Participants) | 3 | 0 | 1 | 0 | 8 | 5
  HIV VL, Month 3 | 75.00 (37.75) |  | 84.00 (NA) — There were not enough subjects for SD analysis to be computed. |  | 19453.50 (11878.74) | 16270.00 (15785.91)
  HIV VL, Month 6: number analyzed (Participants) | 4 | 1 | 2 | 1 | 7 | 5
  HIV VL, Month 6 | 19699.25 (39272.50) | 112.00 (NA) — There were not enough subjects for SD analysis to be computed. | 66053.50 (93328.90) | 51.00 (NA) — There were not enough subjects for SD analysis to be computed. | 37091.29 (33678.60) | 46429.60 (52567.42)
  HIV VL, Month 7: number analyzed (Participants) | 3 | 4 | 1 | 0 | 7 | 5
  HIV VL, Month 7 | 530.67 (785.50) | 55.75 (6.29) | 248.00 (NA) — There were not enough subjects for SD analysis to be computed. |  | 35534.00 (39549.42) | 25774.60 (27360.66)
  HIV VL, Month 18: number analyzed (Participants) | 3 | 3 | 1 | 0 | 7 | 5
  HIV VL, Month 18 | 70.33 (29.54) | 92.67 (64.53) | 48.00 (NA) — There were not enough subjects for SD analysis to be computed. |  | 60597.00 (48313.15) | 14742.60 (18306.17)

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: within 7 days (Days 0-6) post-vaccination. Unsolicited Adverse Events (AEs): within 30 days (Days 0-29) post-vaccination. Serious Adverse Events (SAEs): during the entire study period (from Month 0 up to Month 18).
Arm/Group | GSK1437173A Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/49
Serious Adverse Events (participants affected / at risk) | 6/74 | 2/49
Other Adverse Events (participants affected / at risk) | 72/74 | 29/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1437173A Group (N=74) | Placebo Group (N=49)
Anal abscess (Infections and infestations) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Laryngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK1437173A Group (N=74) | Placebo Group (N=49)
Pain (General disorders) | 72/73 | 6/48 — This solicited local symptom was only collected from those subjects who had their symptom sheets filled in.
Redness (General disorders) | 28/73 | 0/48 — This solicited local symptom was only collected from those subjects who had their symptom sheets filled in.
Swelling (General disorders) | 20/73 | 0/48 — This solicited local symptom was only collected from those subjects who had their symptom sheets filled in.
Fatigue (General disorders) | 55/73 | 14/48 — This solicited general symptom was only collected from those subjects who had their symptom sheets filled in.
Gastrointestinal (General disorders) | 28/73 | 11/48 — This solicited general symptom was only collected from those subjects who had their symptom sheets filled in.
Headache (General disorders) | 47/73 | 15/48 — This solicited general symptom was only collected from those subjects who had their symptom sheets filled in.
Myalgia (General disorders) | 54/73 | 9/48 — This solicited general symptom was only collected from those subjects who had their symptom sheets filled in.
Shivering (General disorders) | 37/73 | 5/48 — This solicited general symptom was only collected from those subjects who had their symptom sheets filled in.
Temperature (General disorders) | 22/73 | 3/48 — This solicited general symptom was only collected from those subjects who had their symptom sheets filled in.
Influenza like illness (General disorders) | 6 | 1
Nasopharyngitis (Infections and infestations) | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.